CLINICAL TRIAL: NCT01476202
Title: A Pilot Study to Evaluate Relief of Provoked Acute Craving by Nicotine Mouth Strip, Nicorette ® Nicotine Lozenge and Gum
Brief Title: Provoked Craving Relief Study by NRT
Acronym: NRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2111378
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2012-04

CONDITIONS: Smoking Cessation
Keywords: craving, provoked craving, smoking cessation, nicotine replacement therapy, NRT
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nicotine mouth strip (Experimental): single dose
  Interventions: Drug: nicotine
- nicotine lozenge (Active Comparator): single dose
  Interventions: Drug: nicotine
- nicotine gum (Active Comparator): single dose
  Interventions: Drug: nicotine

INTERVENTIONS:
Drug: nicotine — nicotine in the form of a mouth strip, lozenge and gum

SUMMARY:
This study is designed to assess the ability of the mint nicotine mouth strip to relieve provoked cigarette craving in light smokers compared to nicotine lozenge and nicotine gum.

ELIGIBILITY:
Inclusion Criteria:

* Smoking Status: Current cigarette smokers who have smoked regularly for at least a year and smoke their first cigarette more than 30 minutes after waking up.

Exclusion Criteria:

* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to nicotine (or closely related compounds) or any of the stated ingredients in formulation.
* Prior Concomitant Medication: a. Treatment with known enzyme altering agents (e.g. carbamazepine, phenytoin, cimetidine, sodium valporate) within 30 days of the craving provocation visit. b. Use of any prescription psychoactive medication (such as but not limited to antidepressants, antipsychotics, anxiolytics) within 14 days of the craving provocation visit. c. Use of any over-the-counter (OTC) medication that affects central nervous system such as antihistamines, sedating agents, or any compound that would have a sedating effect within 24 hours of the craving provocation visit. d. Use of any nicotine replacement therapy or any other treatment for smoking cessation (e.g. bupropion or varenicline) within one month of screening visit. e. Use of any nicotine containing products at any time during the Provocation/Treatment visit. f. Use of any medications noted in the exclusion criteria, or use of any product that would, in the opinion of the investigator, jeopardize the safety of the subject or impact on the validity of the study results.
* Any disease that, in the opinion of the investigator, may interfere with the absorption, metabolism or excretion of the study product. A medical history that, in the opinion of the investigator, might jeopardise the safety of the subject or the validity of the study results. For example, recent myocardial infarction or cerebrovascular accident (within 12 weeks of the screening visit), phenylketonuria, unstable or worsening angina pectoris, Prinzmetals angina or severe cardiac arrhythmia.
* Expired Carbon Monoxide (CO): Any subject whose CO level rises during the sequestration period (i.e., the subject's expired CO assessments immediately prior to the provoked craving paradigm are higher than the mean baseline CO assessment) and, in the opinion of the investigator, may have smoked during that time.
* Alcohol: Consumption of any alcoholic beverage within 24 hours of the craving provocation visit, as indicated by a positive breath alcohol test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Central Kentucky Research Associates, Inc., Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 140 screened participants, 120 were randomized while 17 participants were screen failures, and 3 participants were not randomized due to other reasons.
Groups:
- Nicotine Mouth Strip 2.5 Milligram (mg): Participants self administered a single dose of 2.5 mg nicotine mouth strip.
- Nicotine Lozenge 2 mg: Participants self administered a single dose of 2 mg nicotine lozenge.
- Nicotine Gum 2 mg: Participants self administered a single dose of 2 mg nicotine gum.
Period: Overall Study
Arm/Group | Nicotine Mouth Strip 2.5 Milligram (mg) | Nicotine Lozenge 2 mg | Nicotine Gum 2 mg
Started | 40 | 40 | 40
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Mouth Strip 2.5 mg: Participants self administered a single dose of 2.5 mg nicotine mouth strip.
- Nicotine Gum 2 mg: Participants self administered a single dose of 2 mg nicotine lozenge.
- Total: Total of all reporting groups
Arm/Group | Nicotine Mouth Strip 2.5 mg | Nicotine Lozenge 2 mg | Nicotine Gum 2 mg | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (11.4) | 34.8 (10.9) | 37.4 (11.5) | 35.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 27 | 72
  Male | 18 | 17 | 13 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Nicotine Craving Score on a VAS
Description: Participants completed a nicotine craving assessment consisting of following five items: I have a desire for a cigarette right now, if it were possible I would smoke right now, All I want right now is a cigarette, I have an urge for a cigarette, I crave a cigarette right now. All participants indicated their craving intensity on a pre-drawn 100 mm scale ranging from 0 (disagree) to 100 (agree). At the end of the craving assessment period, mean VAS score was measured.
Time Frame: Baseline, 50 seconds, 3, 5, 7, 10, 15, 20, 25 and 30 minutes post treatment administration
Population: Intent to Treat (ITT) Population: All randomized participants who had at least one dose of medication and provided at least one craving assessment measurement on treatment. The imputation of missing craving score was based on last observation carried forward (LOCF) technique.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nicotine Mouth Strip 2.5 mg | Nicotine Lozenge 2 mg | Nicotine Gum 2 mg
Number analyzed (Participants) | 40 | 40 | 40
Score on a scale
  50 seconds | -11.3 (17.2) | -1.7 (6.0) | -4.6 (9.0)
  3 minutes | -28.2 (28.8) | -12.0 (20.7) | -17.6 (18.4)
  5 minutes | -35.8 (31.0) | -18.3 (22.8) | -27.2 (24.0)
  7 minutes | -39.0 (33.2) | -25.5 (27.2) | -33.8 (27.5)
  10 minutes | -43.9 (31.8) | -30.0 (26.0) | -38.4 (29.9)
  15 minutes | -45.2 (33.3) | -34.4 (29.1) | -40.2 (30.7)
  20 minutes | -47.9 (30.0) | -37.4 (30.1) | -42.7 (31.6)
  25 minutes | -47.3 (33.8) | -40.7 (30.9) | -43.5 (29.7)
  30 minutes | -45.2 (35.3) | -42.8 (32.1) | -42.3 (31.0)

2. Secondary Outcome: Log Transformed Area Under the Curve of Nicotine Craving Score (AUC)
Description: AUC between the baseline (pre-dose) and the time of measurement of craving on-treatment was determined.
Time Frame: Baseline, 50 seconds, 3, 5, 7, 10, 15, 20, 25, and 30 minutes post treatment administration
Population: Intent to Treat (ITT) Population: All randomized participants who had at least one dose of medication and provided at least one craving assessment measurement on treatment. The imputation of missing craving score was based on LOCF technique.
Measure: Log Mean (95% Confidence Interval); unit: Score on a scale*minutes
Groups:
- Nicotine Mouth Strip 2.5 Milligram (mg): Participants self administered single dose of 2.5 mg nicotine mouth strip.
- Nicotine Lozenge 2 mg: Participants self administered single dose of 2 mg nicotine lozenge.
- Nicotine Gum 2 mg: Participants self administered single dose of 2 mg nicotine gum.
Arm/Group | Nicotine Mouth Strip 2.5 Milligram (mg) | Nicotine Lozenge 2 mg | Nicotine Gum 2 mg
Number analyzed (Participants) | 40 | 40 | 40
Score on a scale*minutes
  AUC (0-50 seconds) | 4.0 [3.99 to 4.05] | 4.1 [4.05 to 4.12] | 4.1 [4.03 to 4.10]
  AUC (0-3 minutes) | 5.1 [5.06 to 5.20] | 5.3 [5.23 to 5.38] | 5.2 [5.17 to 5.32]
  AUC (0-5 minutes) | 5.5 [5.42 to 5.61] | 5.7 [5.65 to 5.84] | 5.7 [5.57 to 5.76]
  AUC (0-7 minutes) | 5.8 [5.64 to 5.87] | 6.0 [5.89 to 6.12] | 5.9 [5.81 to 6.03]
  AUC (0-10 minutes) | 6.0 [5.88 to 6.14] | 6.3 [6.14 to 6.41] | 6.2 [6.05 to 6.31]
  AUC (0-15 minutes) | 6.3 [6.15 to 6.45] | 6.6 [6.42 to 6.73] | 6.5 [6.32 to 6.62]
  AUC (0-20 minutes) | 6.5 [6.35 to 6.68] | 6.8 [6.62 to 6.95] | 6.7 [6.50 to 6.83]
  AUC (0-25 minutes) | 6.7 [6.51 to 6.87] | 6.9 [6.76 to 7.12] | 6.8 [6.64 to 7.00]
  AUC (0-30 minutes) | 6.8 [6.65 to 7.03] | 7.1 [6.87 to 7.25] | 7.0 [6.76 to 7.14]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the smoking abstinence sequestration period and until 5 days following last administration of the investigational product.
Groups:
- Nicotine Mouth Strip 2.5 mg: Participants self administered single dose of 2.5 mg nicotine mouth strip.
Arm/Group | Nicotine Mouth Strip 2.5 mg | Nicotine Lozenge 2 mg | Nicotine Gum 2 mg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 4/40 | 0/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Mouth Strip 2.5 mg (N=40) | Nicotine Lozenge 2 mg (N=40) | Nicotine Gum 2 mg (N=40)
Nausae (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.